CLINICAL TRIAL: NCT07401615
Title: Stereotactic Body Radiotherapy (SBRT) for Reirradiation of Inoperable Lung Lesions: an Italian Multicenter Retrospective Analysis (STRILL IT)
Brief Title: Stereotactic Body Radiotherapy (SBRT) for Reirradiation of Inoperable Lung Lesions
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: STRILL IT
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer; Pulmonary Stereotactic Radiotherapy
Keywords: non small cell lung cancer; pulmonary stereotactic radiotherapy; sbrt; re-irradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- re-irradiation SBRT: Patients treated with re-irradiation SBRT on non small cell lung carcinoma

SUMMARY:
Radiotherapy (radiation treatment) is often used to treat lung cancers and lung tumors that have spread from other cancers. It can be very effective, especially in early-stage lung cancer or when there are only a few tumor sites. Even so, some patients later develop a local recurrence, meaning the cancer comes back in the same area that was previously treated with radiation.

When this happens, treatment options are limited. Surgery can sometimes remove the recurrent tumor, but many patients are not able to have surgery because of their general health or because the tumor is difficult to remove. For these patients, a second course of radiotherapy (called re-irradiation) may be the only possible treatment. One type of radiotherapy, called stereotactic body radiotherapy (SBRT), delivers very high doses of radiation very precisely. SBRT has been used successfully as a second treatment after standard radiotherapy in some patients. However, there is very little information about using SBRT again in patients who already received SBRT the first time.

Because only small studies have been done and the patients were very different from each other, doctors still do not know enough about how safe and effective a second SBRT treatment is. In particular, it is still unclear whether giving another high-dose radiation treatment is possible without causing serious side effects. More research is needed to better understand this option and help guide treatment decisions for patients.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable primary non-small cell lung cancer or other metastatic primaries with lung metastases, already treated with radical dose SBRT
* Inoperable local recurrence (defined as a tumor recurrence overlapping the 50% isodose field) confirmed by documented radiographic findings and/or pathological biopsies within the thoracic area
* Patients had previously received curative intent SBRT with a biologically equivalent dose equal or higher than 75 Gy
* Stereotactic reirradiation with ablative purposes up to 8 fractions
* No active distant metastasis or controlled distant metastasis at the time of re-irradiation
* More than 12 months from previous SBRT
* PS ≤ 2

Exclusion Criteria:

* Previous conventional RT
* Reirradiation with palliative doses
* Reirradiation with conventionally fractionated or mildly hypofractionated RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with Pulmonary stereotactic radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | from treatment to 1 years follow up
  evaluation of treatment safety through toxicities according to the CACTE scale

SECONDARY OUTCOMES:
Number of partecipant with local control | from enrollment to 1 years follow up
  defined as the absence of progression within the field of SABR, assessed by contrast-enhanced CT scan
Time to new systemic treatment | from enrollment to 1 years follow up
  time from the first day of SBRT to change or starting of new systemic therapies
Progression free survival | from enrollment to 1 years follow up
  time from the first day of SABR until the date of detection of progressive disease (in-field or out-field) or death, whichever occurred first.
Overall survival | from enrollment to 1 years follow up
  time from the first day of SABR to death. Patients lost to follow-up have their OS censored at the last date they were known to be alive
Dosimetric parameters related to treatment toxicity | from enrollment to 1 years follow up
  analysis between correlation between treatment dosage and occurrence of toxicity

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - AST Papa Giovanni XXIII, Bergamo, Bergamo
  - Radiotherapy Department, Ospedale Bellaria Carlo Alberto Pizzardi, Bologna, Bologna
  - REM Radioterapia, Catania, Catania
  - Radiation oncology unit, Ospedale San Raffaele, Milan, Milano
  - Radiotherapy Department, Istituto Europeo di Oncologia, Milan, Milano
  - IRCCS Humanitas Research Hospital, Rozzano, Milano
  - Radiotherapy Department, IRCCS Istituto Nazionale Fondazione G. Pascale, Napoli, Napoli
  - Centro Fondazione Policlinico Universitario "A. Gemelli", Radioterapia Oncologica, Roma, Roma
  - Radioterapia Oncologica - Ospedale dell'Angelo, Venezia, Venezia
  - Advanced Radiation Oncology Department, IRCCS Sacro Cuore Don Calabria Hospital, Cancer Care Center, Negrar, Verona
  - AOUI Verona, DAI Chirurgia e Oncologia - Radioterapia Oncologica, Verona, Verona

IPD SHARING:
Plan to Share IPD: No